CLINICAL TRIAL: NCT06435468
Title: Biocollection for the Study of Genetic and Immunological Abnormalities in Rare Pediatric-onset Autoimmune and Auto Inflammatory Diseases
Brief Title: Biocollection of Rare Pediatric-onset of Autoimmune and Autoinflammatory Diseases
Acronym: GENIALII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_1252
Record Dates: First submitted 2024-05-07; First posted 2024-05-30 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus; Autoimmune Diseases; Autoinflammatory Disease; Genetic Disease
Keywords: Systemic Lupus; Genetic; rare autoimmune disease; rare autoinflammatory diseases; Pediatric-onset disease
MeSH Terms: conditions — Autoimmune Diseases; Genetic Diseases, Inborn | interventions — Blood Specimen Collection; Genetic Testing

STUDY DESIGN:
Intervention Model Description: prospective, multicenter, national study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with with a rare dysimmune disease (Experimental): minors or adults of any age with a rare dysimmune disease characterized by autoimmunity, autoinflammation or early lymphoproliferation, with onset in childhood (<18 years), or syndromic or familial.
  Interventions: Genetic: Blood sample for genetic analysis; Other: Blood sample for immunological response assessments; Other: Blood sample to identify relevant biomarker of the disease
- Healthy volunteer participants (Other): minor or adult participant without age restriction weighing more than 5 kg
  Interventions: Other: Blood sample for immunological response assessments; Other: Blood sample to identify relevant biomarker of the disease

INTERVENTIONS:
Genetic: Blood sample for genetic analysis — genetic analysis (WES, WGS) for the identification of germline and somatic mutations responsible for rare autoimmune diseases or auto-inflammatory pathologies (pediatric or syndromic or familial) that began in childhood
  Arms: Patient with with a rare dysimmune disease
Other: Blood sample for immunological response assessments — Identifying specific immunological factors in patients with rare pediatric autoimmune and auto inflammatory diseases
Other: Blood sample to identify relevant biomarker of the disease — Research biomarkers for diagnosis, prognosis and monitoring of disease activity

SUMMARY:
Rare diseases are defined as those that affect one person in 2,000, or around three million people in France. The majority of rare diseases are caused by genetics and tend to be severe when they begin in childhood. Autoimmune and autoinflammatory diseases, such as systemic lupus, juvenile dermatomyositis, and juvenile idiopathic arthritis, are examples of rare pediatric diseases. While autoimmune diseases are characterized by an inappropriate adaptive immune response, autoinflammatory diseases involve an excess of the innate immune response. The precise mechanisms of these diseases are not yet fully understood, but recent research has led to advances in their diagnosis and identification, particularly in early onset and familial forms. However, the rarity of these diseases and limited availability of biological samples pose significant challenges.

This study aims to create a biological collection, which includes primary cells (PBMC), DNA, RNA, lymphoblastic lines, and serum, that will help identify genetic and immunological abnormalities in rare autoimmune and autoinflammatory diseases through various research projects.

DETAILED DESCRIPTION:
A disease is said to be "rare" when it affects one person in 2,000, which represents three million people in France. Most rare diseases (80%) are genetic in origin ; the earlier they start in childhood, the more severe they can be. Rare pediatric diseases include autoimmune diseases (systemic lupus, juvenile dermatomyositis and juvenile idiopathic arthritis) and autoimmune diseases (interferonopathies, FMF, CAPS, TRAPS, and DADA2). Systemic autoimmune diseases are characterized by an inappropriate adaptive immune response (mediated by autoreactive T and/or B lymphocytes) with the production of autoantibodies directed against the constituents of the self (tolerance breakdown). Autoinflammatory diseases, unlike autoimmune diseases, correspond to an excess in the innate immune response (cytokines, macrophages, NK cells, granulocytes, etc.)..The precise pathophysiological mechanisms of these diseases have yet to be fully elucidated. Recent research has led to advances in the diagnosis and identification of monogenic forms of these diseases, particularly in early onset, familial, and syndromic forms. Nevertheless, the rarity of these diseases and limited availability of biological samples are major challenges that need to be overcome.

Thus, the aims of this study were as follows:

- The creation of a biological collection: primary cells (PBMC), DNA, RNA, lymphoblastic lines, and serum, which, through various research projects, will help identify genetic and immunological abnormalities in rare autoimmune and autoinflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients
* minor or adult patient of any age with a rare dysimmune disease characterized by autoimmunity or auto-inflammation or early lymphoproliferation, having started in childhood (<18 years), or syndromic or familial
* relative of a minor or adult patient with a rare dysimmune disease characterized by autoimmunity or auto-inflammation or early lymphoproliferation, having started in childhood (<18 years of age) or syndromic or familial,
* weight greater than 5 kg
* Patient/parents/guardians who were informed of the study and signed the consent form.
* patient affiliated to a social security scheme

Healthy volunteer participants

* minor or adult participants with no age restrictions
* weight over 5 kg
* Subject /Parents/guardians who were informed of the study and signed a consent form.
* Patient affiliated to a social security scheme

Exclusion Criteria:

Patients

- Subjects /Parents/guardians, refusing to participate in the study

Healthy volunteer participants :

* active infection (viral, bacterial, parasitic)
* history of neoplasia (< 5 years) or current neoplasia
* participants with a personal or family history of autoimmune disease
* immunocompromised participant (immune deficiency or transplant recipient)
* Subjects/parents/guardians refusing to participate in the study
* Adults under legal protection (guardianship, curatorship)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2035-02-27 (Estimated); Study Completion 2035-07-27 (Estimated)

PRIMARY OUTCOMES:
To Identify germline and somatic mutations responsible for rare autoimmune diseases or auto-inflammatory pathologies (pediatric or syndromic or familial) that began in childhood | Baseline
  Identification of germline or somatic genetic mutations, based on high-throughput sequencing data (exome, genome or transcriptome).

SECONDARY OUTCOMES:
Measurement of disease activity according to Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | Baseline
  score (Min value: 0 - Max value: 105), with higher values mean higher disease activity
Levels of anti-double stranded DNA | Baseline
  in patients sera
Levels of complement components C3 and C4 | Baseline
  in patients sera
Level of IFN Signature score | Baseline
  Mesured by 6-gene Type 1 IFN Signature Score
Concentration of circulating IFN-alpha | Baseline
  In serum using single-molecule array digital ELISA technology (Simoa)
Presence or absence of anti-type I interferons autoantibodies | Baseline
  in patients sera

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Service de rhumatologie pédiatrique Hôpital Femme-Mère-enfant, Bron, Bron
  - Hôpital Jeanne de Flandre (CHU de Lille), Lille, Lille
  - Hôpital Claude Huriez (CHU de Lille), Lille, Lille
  - Hôpital Archet 2, Nice, Nice
  - Hôpital Necker-Enfants Malades (AP-HP), Paris, Paris
  - Hôpital Robert Debré (AP-HP), Paris, Paris
  - Hôpital Kremlin-Bicêtre (AP-HP), Paris, Paris
  - Hôpital Nord (CHU ST-Etienne), Saint-Etienne, Saint Etienne
  - Hôpital Couple Enfant, Grenoble
  - Dr Isabelle MELKI, Paris
  - CLCC Henri Becquerel, Rouen
  - Pr Ariane ZALOSZYC, Strasbourg
  - Dr Vanessa Remy-Piccolo, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No